CLINICAL TRIAL: NCT06916299
Title: Short-term Stability of Tooth-borne vs Bone-borne Maxillary Expansion: A Parallel Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Michele Cassetta, Full Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: URomLS_5951relapse
Record Dates: First submitted 2025-03-20; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Orthodontic Appliance; Orthodontic Appliances; Orthodontic Relapse
Keywords: relapse; stability; miniscrews; rapid maxillary expansion
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tooth borne expansion (Active Comparator)
  Interventions: Diagnostic Test: dental casts; Device: tooth-borne expander insertion
- bone-borne expansion (Experimental)
  Interventions: Diagnostic Test: dental casts; Procedure: miniscrew and bone-borne expander insertion

INTERVENTIONS:
Diagnostic Test: dental casts — At the end of the planned expansion, an 8-month retention period was expected. At this time, the expansion device was removed, and impressions were taken in both groups (T1).
  At 12-month follow-up (T2), new impressions were taken in both groups to evaluate, at dental level, the relapse in the short term. Fig 1
Device: tooth-borne expander insertion — tooth-borne expander delivery.
  Arms: tooth borne expansion
Procedure: miniscrew and bone-borne expander insertion — Insertion of the paramedian miniscrews in a totally guided procedure, and after was delivered the tooth-borne expander
  Arms: bone-borne expansion

SUMMARY:
This prospective parallel cohort study aimed to compare the short-term stability of maxillary expansion achieved with tooth-borne (Hyrax) and bone-borne expanders.

A total of 36 patients (mean age: 12.3 ± 0.6 years) with transverse maxillary deficiency (≥8 mm) were randomly assigned to two groups: Group A (tooth-borne Hyrax) and Group B (bone-borne expander with four mini-screws). Both groups followed the same activation protocol and underwent an 8-month retention period. After this period, the expansion devices were removed, and relapse was assessed at 12 months post-expansion (T2), corresponding to 4 months after device removal. Digital dental models were analyzed using linear measurements, and statistical analysis was conducted using t-tests (p ≤ 0.05).

DETAILED DESCRIPTION:
The present prospective study aimed to compare, through a parallel cohort study, the stability of the results obtained at the dental level of tooth-borne (hyrax) and bone-borne maxillary expansion.

It has been hypothesized that some degree of post-treatment relapse is always present and that there are no significant differences between the two types of RME.

The clinical investigation was conducted following the ethical principles of the World Medical Association Declaration of Helsinki. The parents or guardians were informed of the content, risks, and benefits of the study, and written consent was obtained. The local ethics committee approved the investigation (Rif. N. 5951- Prot. N. 250/2020). Of the 200 eligible subjects, 26 were included. The patients were randomly divided into two groups, Group A and Group B, using the statistical software Clinstat (Martin Bland, York, UK). Group A was treated with a tooth-borne hyrax expander, with two bands placed on the first permanent molars. Group B was treated with a bone-borne expander supported by four mini-screws, two inserted in the paramedian position and two in the parapalatal position. The mini-screws were placed using a computer-guided technique, assisted by a surgical guide (Easy Driver; Uniontech Orthodontic Lab, Parma, Italy), created with a 3D printer (Stratasys OrhoDesktop; Stratasys, Rehovot, Israel). The insertion site, angle, length, and diameter of the miniscrews were planned using specialized software that matched CBCT images with STL files of the digital dental models. Both the mini-screws (Benefit system; PSM Medical Solutions, Tuttlingen, Germany) and the expansion devices were inserted in the same session. In both groups, the same expansion screw (10 mm; hyrax click; Dentaurum, Ispringen, Germany) and the same activation protocol were used: 4 turns on the first day, followed by 3 turns per day for the next twelve days. An 8 mm screw opening (0.2 mm per turn) was achieved in both groups. At the end of the planned expansion, an 8-month retention period was expected. At this time, the expansion device was removed, and impressions were taken in both groups (T1).

At 12-month follow-up (T2), new impressions were taken in both groups to evaluate, at dental level, the relapse in the short term. Fig 1 The plaster study models deriving from the impressions taken at T1 and T2 were scanned using a 3D scanner (Raptor3DX platform VYLO) and saved as stereolithographic files (STL). The measurements on the three-dimensional models were carried out by two operators (M.M. and R.G.) using dedicated software (Exocad DentalDB 3.1 Rijeka 8349 Version 3.1) and repeated one month later to evaluate the intra-operator and inter-operator variability. Statistical analysis Data were collected on an Excel database (Microsoft, Redmond, WA, USA) and analysed using statistical analysis software (Python 3.6). Descriptive statistical analysis (mean values and standard deviation) was performed to evaluate the relapse at twelve months (T2), after four months since the device was permanently removed.

The measurements on the eight-month and twelve-month models (ΔT2-T1) were performed, and the T-test was used to analyse the differences between the two groups.

Cohen's kappa coefficient (k) was used to evaluate the interobserver variability. Intraclass correlation coefficient was used to assess the intra-observer variability.

In all analyses, a P ≤0.05 was considered as an indicator of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian children in late mixed dentition or permanent dentition,
* unilateral or bilateral transverse maxillary deficiency of at least 8 mm,
* no patients with skeletal Class III and/or open bite,
* no previous orthodontic treatment,
* good oral hygiene,
* good quality of the plaster models to allow a suitable scanning.

Exclusion Criteria:

* systemic syndrome involved

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
stability | up to 14 months
  Variable Description MV Distance between the mesio-vestibular cusps of the upper first permanent molars.
  MP Distance between the mesio-palatal cusps of the upper first permanent molars.
  CP Distance between the central pits of the upper first permanent molars. AC Distance between the most vestibular points of the buccal alveolar crest at the level of the dental neck of the upper first permanent molars.
  VP Distance between the most vestibular points of the mesial vestibular cusps of the upper first permanent molars.
  ALright Right maxillary arch length, evaluated as the distance between the mesial contact point of the upper right first permanent molar and the contact point between the upper central incisors.
  ALleft Left maxillary arch length, evaluated as the distance between the mesial contact point of the upper left first permanent molar and the contact point between the upper central incisors.
  AP The arch perimeter was evaluated as the addition of the length of the segments A(1.4-1.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Sciences, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No